CLINICAL TRIAL: NCT01945827
Title: Evaluation of DeltaMaxx® Microcoil System in Intracranial Aneurysms
Status: Withdrawn | Type: Observational
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Other Study IDs: CD-000036-PRO
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DeltaMaxx treated Patients
  Interventions: Device: DeltaMaxx Microcoil System

INTERVENTIONS:
Device: DeltaMaxx Microcoil System

SUMMARY:
The primary objective of this registry is to assess the safety and angiographic outcomes of endovascular treatment of intracranial aneurysms using the DeltaMaxx Microcoil System.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥18 and ≤80 with a diagnosis of ruptured or unruptured intracranial aneurysm judged suitable for selective endovascular treatment by coil occlusion during single procedure
* Investigator intends to use DeltaMaxx Microcoil system during coiling procedure
* Investigator intends to use only Codman Neuro microcoils during coiling procedure
* Aneurysm size [largest measurement from the cross sectional images to determine overall aneurysm size, not just the lumen] ≥6 mm
* If ruptured aneurysm: Hunt and Hess 1, 2, or 3
* If unruptured aneurysm: Subject grade Modified Rankin Scale 0 - 2
* The subject or his/her Legally Authorized Representative must voluntarily provide Informed Consent for participation in this study and agree to return for all study visits.

Exclusion Criteria:

* Prior treatment (surgical or endovascular) of the target aneurysm
* Subjects with more than one aneurysm (>2 mm) that have been treated with endovascular or clipping techniques in the past 30 days.
* Subject with social, medical or psychological conditions that interfere with treatment and follow-up evaluation
* Women who are pregnant or plan to become pregnant during the study
* Life expectancy less than 12 months.
* Presence of arteriovenous malformation
* Fusiform, mycotic, traumatic, or tumoral aneurysms
* Planned aneurysm treatment by parent vessel occlusion
* Subject enrolled in any concurrent study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been diagnosed with a ≥ 6 mm intracranial aneurysm.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Objective - Angiographic Outcomes | 12 Months
  The Primary Effectiveness endpoint is the immediate post-procedure and 12-month angiographic occlusion rates assessed by the independent core lab using the modified Raymond-Roy Grading Scale (RRGS) scale
Primary Safety Endpoint - Neurological Morbidity and Mortality | 12 months
  Neurological Morbidity and Mortality as determined by the NIH Stroke Scale and all-cause mortality, regardless of relationship to the treatment, will be captured over the course of the study

SECONDARY OUTCOMES:
Packing Density | 24 hours
  Packing density as measured by volumetric filling of the aneurysm post-procedure after the coils have been placed as indicated by angiographic films taken at the end of the coiling procedure
Recurrence Rate | 12 months
Re-treatment Rate | 12 months